CLINICAL TRIAL: NCT05646797
Title: A Phase 1/1b Study of ASP2074 in Participants With Metastatic or Locally Advanced Solid Tumors
Brief Title: A Study of ASP2074 in Adults With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company Strategic Reasons
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2074-CL-0101; jRCT2031220554 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
Keywords: Solid Tumor;; Malignancy;; Metastasis;; cancer;; ASP2074;; Pharmacokinetics
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ASP2074 Dose Escalation (Part 1) (Experimental): Participants will be assigned to sequentially or in parallel escalating dose/regimen cohorts of ASP2074 in three parts (Part A, B and C). Part B and Part C will be opened sequentially based upon sponsor review of emerging data.
  Interventions: Drug: ASP2074
- ASP2074 Dose Expansion (Part 2) Colorectal Adenocarcinoma (Experimental): Participants will receive ASP2074 with dose/regimen selected from dose escalation (Part 1).
  Interventions: Drug: ASP2074
- ASP2074 Dose Expansion (Part 2) Esophageal or GEJ Adenocarcinoma (Experimental): Participants will receive ASP2074 with dose/regimen selected from dose escalation (Part 1).
  Interventions: Drug: ASP2074
- ASP2074 Dose Expansion (Part 2) Pancreatic Adenocarcinoma (Experimental): Participants will receive ASP2074 with dose/regimen selected from dose escalation (Part 1).
  Interventions: Drug: ASP2074

INTERVENTIONS:
Drug: ASP2074 — intravenous (IV) infusion

SUMMARY:
ASP2074 is a potential new treatment for people with certain solid tumors. Before ASP2074 is available as a treatment, the researchers need to understand how it is processed by and acts upon the body. This information will help find a suitable dose and check for potential medical problems from the treatment. People in this study will be adults with metastatic or locally advanced solid tumors. Metastatic means the cancer has spread to other parts of the body. They will have been previously treated with all available standard therapies and they may no longer be benefitting from further treatment.

There are 2 main aims of this study. The first is to learn if people with certain solid tumors have any medical problems after receiving different doses of ASP2074. The second is to find a suitable dose of ASP2074 to use in future studies.

This study will be in 2 parts.

In Part 1, different small groups of people will receive lower or higher doses of ASP2074. Any medical problems will be recorded at each dose. This is done to find suitable doses of ASP2074 to use in Part 2 of the study. The first group will receive the lowest dose of ASP2074. A medical expert panel will check the results from this group and decide if the next group can receive a higher dose of ASP2074. The panel will do this for each group until all groups have taken ASP2074 or until suitable doses have been selected for Part 2.

In Part 2, other different small groups of people will receive ASP2074 with the most suitable doses worked out from Part 1. This will help find a more accurate dose of ASP2074 to use in future studies.

ASP2074 will be given as an infusion on the first day of each treatment cycle. The people in this study will have treatment cycles until: they have medical problems from the treatment; their cancer gets worse; they start other cancer treatment; they ask to stop treatment; or they do not come back for treatment.

People will visit the clinic on certain days during their treatment, with extra visits during the first 2 cycles of treatment. During these visits, the study doctors will check for any medical problems from ASP2074. At some visits, other checks will include a medical examination, laboratory tests and vital signs. Vital signs include temperature, pulse, and blood pressure. Also, blood and urine samples will be taken. Electrocardiograms will be done to check the heart rhythm during the study. Tumor samples will be taken during certain visits before treatment begins, during treatment, and when treatment has finished.

People will visit the clinic within 7 days after stopping treatment. The study doctors will check for any medical problems from ASP2074. Other checks will include a medical examination, laboratory tests and vital signs. Then, people may visit the clinic at 30 days after stopping treatment. Thirty and 90 days after the last dose, the study doctors will check for any medical problems from ASP2074. People will have their vital signs checked and have some laboratory tests. After this, people will continue to visit the clinic every 6 weeks. This is to check the condition of their cancer. They will do this until their cancer is worse, they start other cancer treatment, they ask to leave the study, or they do not come back for treatment. Then, the study doctors will call every 12 weeks for up to 1 year or until that person asks to leave the study, the study is stopped, or the person cannot be reached.

ELIGIBILITY:
Inclusion Criteria:

* Participant has locally-advanced (unresectable) or metastatic solid tumor malignancy (no limit to the number of prior treatment regimens) which is confirmed by available pathology records or current biopsy. For dose escalation, the participant must have colorectal, pancreatic, gastric cancer, esophageal or Gastroesophageal junction (GEJ) adenocarcinoma. For the tumor-specific expansion cohorts, the participant must have colorectal adenocarcinoma, esophageal or GEJ adenocarcinoma, or pancreatic adenocarcinoma.
* Participant has at least 1 measurable lesion per RECIST v1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant has progressed or failed to tolerate after receiving all standard approved therapies or is no longer eligible for standard therapy (no limit to the number of prior treatment regimens).
* Participant has an Eastern Cooperative Oncology Group (ECOG) Status of 0 or 1.
* Participants who have received radiotherapy must have completed this therapy (including stereotactic radiosurgery) at least 2 weeks prior to study intervention administration.
* Participant's adverse events (excluding alopecia) from prior therapy have improved to grade 1 or baseline for the participant (e.g., grade 2 hypothyroidism) within 14 days prior to the first dose of study intervention.
* Participant has predicted life expectancy >/= 12 weeks.
* Participant must meet all of the criteria based on laboratory tests. In case of multiple laboratory data within this period, the most recent data should be used. If a participant has received a recent blood transfusion, the laboratory tests must be obtained >/= 2 weeks after any blood transfusion.
* Female participant is not pregnant confirmed by serum pregnancy test and medical evaluation by interview and at least 1 of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP)
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 90 days after final study intervention administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 90 days after final study intervention administration.
* Female participant must not donate ova starting at first dose of study intervention and throughout the study period and for 90 days after final study intervention administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 90 days after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 90 days after final study intervention administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 90 days after final study intervention administration.
* Participant agrees not to participate in another interventional study while receiving study treatment in the present study.

Exclusion Criteria:

* Participant has received other investigational agents or devices concurrently or within 21 days or 5 half-lives, whichever is shorter, prior to first dose of study intervention administration.
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP2074 or any components of the formulation used.
* Participants with squamous cell colorectal carcinoma; gastrointestinal stromal tumor and neuroendocrine carcinomas.
* Participant weighs < 40 kg.
* Participant requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to study intervention administration. Participants using a physiologic replacement dose of hydrocortisone or its equivalent (defined as up to 30 mg per day of hydrocortisone or up to 10 mg per day prednisone), receiving a single dose of systemic corticosteroids, or receiving systemic corticosteroids as premedication for radiologic imaging contrast use is eligible.
* Participant has symptomatic CNS metastases or participant has evidence of unstable CNS metastases even if asymptomatic (e.g., progression on scans). Participants with previously treated CNS metastases are eligible, if they are clinically stable and have no evidence of central nervous system (CNS) progression by imaging for at least 4 weeks prior to start of study treatment and are not requiring immunosuppressive doses of systemic steroids (> 30 mg per day of hydrocortisone or > 10 mg per day of prednisone or equivalent) for longer than 2 weeks.
* Participant has an active autoimmune disease. Participants with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy, or skin disorders (e.g., vitiligo, psoriasis, or alopecia) not requiring systemic treatment are allowed.
* Participant was discontinued from prior immunomodulatory therapy due to a grade >/= 3 toxicity that was mechanistically related (e.g., immune related) to the agent.
* Participant is known to have HIV infection. However, participants with HIV infection with CD4+ T-cell counts ≥ 350 cells/μL and no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the past 6 months are eligible. NOTE: Screening for human immunodeficiency virus (HIV) infection should be conducted per local requirements.
* Participant is known to have active hepatitis B (positive hepatitis B surface antigen (HBsAg)) or hepatitis C infection. NOTE: Screening for these infections should be conducted per local requirements.

  * For participant who is negative for HBsAg, but hepatitis B core antibody (HBcAb) positive, a hepatitis B virus (HBV) DNA test will be performed and if positive the participant will be excluded.
  * Participant with positive hepatitis C virus (HCV) serology, but negative HCV RNA test results are eligible.
  * Participant treated for HCV with undetectable viral load results are eligible
* Participant has received a live vaccine against infectious diseases within 28 days prior to initiation of study treatment.
* Participant with a history of interstitial lung disease (ILD) or non-infectious pneumonitis, or currently has ILD/pneumonitis.
* Participant has an infection requiring systemic therapy within 14 days prior to study drug treatment.
* Participant has received a prior allogeneic bone marrow or solid organ transplant.
* Participant is expected to require another form of antineoplastic therapy while on study treatment.
* Participant with a history of the following significant cardiovascular disease will be excluded:

  * Participant has inadequately controlled hypertension on antihypertensive medications.
  * Participant has a history of myocardial infarction or unstable angina within 6 months prior to day 1.
  * Participant has New York Heart Association Class II or greater Congestive heart failure (CHF).
  * History of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to study treatment.
  * Participant has significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study treatment.
  * Participant has cardiac arrhythmia, complete left bundle branch block, obligate use of a cardiac pacemaker, long QT syndrome or right bundle branch block with left anterior hemiblock (bifascicular block).
  * Participant has a corrected time from the start of the Q wave to the end of the T wave (QT) interval (single ECG) using Fridericia's formula (QTcF) > 450 msec during screening. A single 12-lead ECG will be performed during screening.
* Participant has had psychiatric illness/social situations that would limit compliance with study requirements.
* Participant has a prior malignancy, other than the current malignancy for which the participant is seeking treatment, active (i.e., requiring treatment of intervention) within the previous 2 years except for locally curable malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast.
* Participant has had major surgery within 28 days prior to the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) for ASP2074 | Up to up to 28 Days
  A Dose Limiting Toxicity (DLT) is defined as any prespecified Adverse events (AEs) or laboratory findings occurring during the DLT evaluation period excluding toxicities clearly related to disease progression or intercurrent illness.
Number of participants with Adverse Events (AEs) | Up to 15 Months
  Adverse events (AEs) will be coded using MedDRA. An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants with Serious Adverse Events (SAEs) | Up to 15 Months
  A Serious Adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other medically important event.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 13 Months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to 15 Months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to 15 Months
  Number of participants with potentially clinically significant ECG values.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 21 Months
  ORR is defined as is defined as the proportion of participants whose best overall response is a confirmed Complete Response (CR) or Partial Response (PR).
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 21 Months
  ORR is defined as the proportion of participants whose best overall response is a confirmed Complete Response (CR) or Partial Response (PR).
Duration of Response (DOR) per iRECIST | Up to 21 Months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented disease progression (PD) or death due to any cause, whichever occurs first. DOR will only be calculated for participants with confirmed CR or PR.
Duration of Response (DOR) per RECIST v1.1 | Up to 21 Months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented PD or death due to any cause, whichever occurs first. DOR will only be calculated for participants with confirmed CR or PR.
Disease Control Rate (DCR) per iRECIST | Up to 21 Months
  DCR is defined as the proportion of participants whose best overall response is confirmed CR, PR or stable disease (SD).
Disease Control Rate (DCR) per RECIST v1.1 | Up to 21 Months
  DCR is defined as the proportion of participants whose best overall response is confirmed CR, PR or stable disease (SD).
Change from Baseline in Serum CA19-9 levels in participants with pancreatic cancer | Baseline and up to 21 Months
  Serum carbohydrate antigen 19-9 (CA19-9) levels will be recorded in participants with pancreatic cancer.
Pharmacokinetics (PK) of ASP2074 in serum: AUC(0-336h) | Up to 12 Months
  Area under the concentration-time curve from time zero to 336 hours post dose (AUC(0-336h)) will be recorded from the PK serum samples collected.
Pharmacokinetics (PK) of ASP2074 in serum: Cmax | Up to 12 Months
  Maximum concentration (Cmax) will be recorded from the PK serum samples collected.
Pharmacokinetics (PK) of ASP2074 in serum: Ctrough | Up to 12 Months
  Concentration immediately prior to dosing at multiple dosing (Ctrough) will be recorded from the PK serum samples collected.
Pharmacokinetics (PK) of ASP2074 in serum: tmax | Up to 12 Months
  Time of maximum concentration (tmax) will be recorded from the PK serum samples collected.
Change from Baseline in target antigen expression | Baseline and up to Day 40
  Comparison of target antigen expression in baseline versus on-treatment tumor biopsies will be performed.
Change from Baseline in tumor CD8 infiltration/ activation | Baseline and up to Day 40
  Comparison of CD8 infiltration/ activation in baseline versus on-treatment tumor biopsies will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (13):
- United States (8):
  - University of California Davis Health System, Sacramento, California
  - University of Iowa Hospitals, Iowa City, Iowa
  - Karmanos Cancer Institute, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Duke University, Durham, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Next Oncology - Oncology, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Japan (5):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14990&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/2074-CL-0101